CLINICAL TRIAL: NCT05802355
Title: Manual Diaphragmatic Release: Is It Helpful for Cleaning-laborers With Work-related Respiratory Hazards in Overcoming the Upsetting Respiratory Symptoms, Boosting Immune Response, and Enhancing Functional Ability?
Brief Title: Manual Diaphragm Release in Cleaning Laborer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maged Basha (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor-Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Organization: Qassim University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/022/37
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Respiratory System Abnormalities
Keywords: Respiratory hazards; pulmonary function; chest wall mobility; functional ability; Manual Diaphragmatic Release
MeSH Terms: conditions — Respiratory System Abnormalities | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Diaphragm Release (Experimental): received 3sessions/ week for 12 consecutive weeks.
  Interventions: Other: Manual Diaphragm Release
- control group (Experimental): received 3sessions/ week for 12 consecutive weeks.
  Interventions: Other: control group

INTERVENTIONS:
Other: Manual Diaphragm Release — The participant was supine, with his or her limbs relaxed. With the therapist's forearms aligned toward the participant's shoulders, the therapist gradually increased the depth of contact inside the costal margin during the subsequent respiratory cycles.
  Other Names: inspiratory resistance
  Arms: Manual Diaphragm Release
Other: control group — Respiratory re-training was given to participants in control group in form of slow and deep diaphragmatic breathing, exhalation through the nose with pursed lips (the participants were trained to emphasis on expiratory pressure against pursed lips), Breathing control and breathing-hold exercises, and Relaxation techniques:
  Other Names: Respiratory re-training
  Arms: control group

SUMMARY:
This study intended to examine the effect of manual diaphragm release on pulmonary function, chest wall mobility, and functional ability in female occupational cleaners with respiratory hazards.

DETAILED DESCRIPTION:
Cleaning chores have been linked to exposure to various chemical agents that have the potential to cause harmful effects on both the respiratory system and cardiovascular markers, many cleaning products and disinfectants contain ingredients that can act as airway irritants. One of the physical therapy procedures that is used to manage chest disorders is manual diaphragm release which aims to lengthen the diaphragm musculature whereas encouraging better and more proficient contraction.

ELIGIBILITY:
Inclusion Criteria:

* Female occupational cleaners.
* Age between 35 and 45.
* Had work-related respiratory hazards.
* Clinically stable.
* No exacerbation in the previous 6 weeks.
* Working in an occupation with respiratory hazards for at least 2 years.
* Mild to moderate air way obstruction.
* Willingness to participate in this study and provide a consent form.

Exclusion Criteria:

* Other cardiopulmonary diseases.
* Body mass index > 30 kg/ m2.
* Previous thoracic or abdominal surgery.
* Smokers and users of tobacco in any form (chewing, snuffing or water pipe).
* Systemic conditions (e.g., diabetes mellitus, hypertension).
* Sever airway obstructions.
* Inability to perform the required exercises.
* Inability to attend the scheduled sessions.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female occupational cleaners working in an occupation with respiratory hazards for at least 2 years.
Enrollment: 36 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Serum IgE | at first week
  The Organon Teknika Microwell system (Organon Teknika Corp, Boxtel, the Netherlands) and an enzyme-linked immunosorbent test kits, were utilized to assess total serum IgE (IU/mL) at 450 nm.
Serum IgE | after 12 weeks
  The Organon Teknika Microwell system (Organon Teknika Corp, Boxtel, the Netherlands) and an enzyme-linked immunosorbent test kits, were utilized to assess total serum IgE (IU/mL) at 450 nm.
Forced vital capacity | at first week
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards
Forced vital capacity | after 12 weeks
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards
Forced expiratory volume in one second | at first week
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards
Forced expiratory volume in one second | after 12 weeks
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards
pulmonary expiratory flow | at first week
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards
pulmonary expiratory flow | after 12 weeks
  measured using a portable MicroLab spirometer (Vyaire Medical, Mettawa, Illinois) in accordance with current lung function testing standards

SECONDARY OUTCOMES:
Chest wall mobility | at first week
  measured using tape measurement with maximum inspiration and expiration and the difference between them has been recorded in (cm).
Chest wall mobility | after 12 weeks
  measured using tape measurement with maximum inspiration and expiration and the difference between them has been recorded in (cm).
Functional performance | at first week
  Assessed using the 6-minute walk test
Functional performance | after 12 weeks
  Assessed using the 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa azab, PhD, Principal Investigator — Cairo University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Zock JP, Kogevinas M, Sunyer J, Jarvis D, Toren K, Anto JM; European Community Respiratory Health Survey. Asthma characteristics in cleaning workers, workers in other risk jobs and office workers. Eur Respir J. 2002 Sep;20(3):679-85. doi: 10.1183/09031936.02.00279702. PMID 12358347
- [Background] Mirabelli MC, London SJ, Charles LE, Pompeii LA, Wagenknecht LE. Occupation and three-year incidence of respiratory symptoms and lung function decline: the ARIC Study. Respir Res. 2012 Mar 20;13(1):24. doi: 10.1186/1465-9921-13-24. PMID 22433119
- [Background] Bruurs ML, van der Giessen LJ, Moed H. The effectiveness of physiotherapy in patients with asthma: a systematic review of the literature. Respir Med. 2013 Apr;107(4):483-94. doi: 10.1016/j.rmed.2012.12.017. Epub 2013 Jan 18. PMID 23333065
- [Result] Malaguti C, Rondelli RR, de Souza LM, Domingues M, Dal Corso S. Reliability of chest wall mobility and its correlation with pulmonary function in patients with chronic obstructive pulmonary disease. Respir Care. 2009 Dec;54(12):1703-11. PMID 19961637
- [Derived] Azab AR, Elnaggar RK, Hamouda DG, Aloraini GS, Alhegaili AS, Ahmed AS, Basha MA, Alsharidah AS, Kamel FH, Elshehawy AA. Respiratory and functional benefits of manual diaphragmatic release for cleaning-laborers exposed to occupational hazards. Physiother Res Int. 2024 Oct;29(4):e70001. doi: 10.1002/pri.70001. PMID 39427332